CLINICAL TRIAL: NCT06698510
Title: Arpraziquantel for Schistosomiasis Control in Preschool-aged Children in Endemic Areas in Kenya and Côte d'Ivoire: A Small-scale Public Health Intervention Study Arpraziquantel for Schistosomiasis Control in Preschool-aged Children in Endemic Areas in Uganda, With Special Consideration of Dose Determination Methods: a Small-scale Public Health Intervention Study in Hoima and Bugiri Districts
Brief Title: Introduction of Arpraziquantel Treatment for Schistosomiasis Control in Preschool-aged Children in Endemic Areas: A Small-scale Public Health Intervention Study
Acronym: ADOPTpilot
Status: Recruiting | Type: Observational
Sponsor: Peter Steinmann (Other)
Collaborators: Technical University Munchen (Unknown); Makerere University (Other); African Institute for Health and Development, Kenya (Unknown); Kenya Medical Research Institute (Other); Kenya Ministry of Health (Other Government); Ministry of Health, Uganda (Other Government); Ministère de la Santé, de l'Hygiène Publique et de la Couverture Maladie Universelle (Unknown); Université Félix Hophouët-Boigny (Unknown); Unlimit Health (Unknown)
Responsible Party: Sponsor-Investigator, Peter Steinmann, Unit Head, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Other Study IDs: 2108p; RIA2019IR-2895; G2020-102 (Other Grant/Funding Number: European and Developing Countries Clinical Trials Partnership (EDCTP); Global Healh Innovative Technology (GHIT) Fund)
Record Dates: First submitted 2024-11-14; First posted 2024-11-21 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Schistosomiasis
Keywords: schistosomiasis; preschool-aged children; praziquantel; arpraziquantel; deworming; pediatric treatment; child health
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- arPZQ distributed through Platform 1 (NTD programmes): Preschool-aged children (24 to 59 months of age) of villages preselected to receive a single oral dose of 50mg/kg or 60mg/kg (depending on country) arpraziquantel as part of the routine schistosomiasis mass drug administration campaigns led by the national NTD programmes.
  Interventions: Drug: Arpraziquantel 150mg dispersible tablet
- arPZQ distributed through Platform 2 (child health days/nutrition programmes): Preschool-aged children (24 to 59 months of age) of villages preselected to receive a single oral dose of 50mg/kg or 60mg/kg (depending on country) arpraziquantel as part of the routine vitamin A distribution/child health days campaigns led by the national nutrition programmes.
  Interventions: Drug: Arpraziquantel 150mg dispersible tablet

INTERVENTIONS:
Drug: Arpraziquantel 150mg dispersible tablet — Arpraziquantel 150mg dispersible tablets given as single oral dose of 50mg/kg (in Kenya and Uganda; for Schistosoma mansoni infection) or 60mg/kg (in Côte d'Ivoire; for mixed infections with S. mansoni / S. haematobium) using weight-based dosing tables as detailed in the summary of product characteristics.

SUMMARY:
The proposed small-scale pilot studies are public health intervention studies implemented through established routine programs and services in the frame of the mass drug administration (MDA) campaigns in Côte d'Ivoire, Kenya and Uganda. In each country two most promising health intervention platforms were selected for pilot distribution of arpraziquantel 150mg (arPZQ).

The aim of the small-scale pilot study is to assess the performance of different platforms for distributing arPZQ, a child-friendly formulation of praziquantel, to the target population (i.e., preschool-aged children (PSAC)) currently missed out in schistosomiasis treatment campaigns.

The specific objectives of the pilot study are:

* To assess the performance of different platforms for delivery of arPZQ to PSAC aged 24 to 59 months in terms of coverage, feasibility and acceptability
* To determine social mobilization and training needs for effective delivery of arPZQ through different platforms

Preventive chemotherapy with arPZQ will be offered systematically to eligible PSAC aged 2 to below 5 years of consenting caregivers resident in the study area and reached through the selected platforms. Adverse events during MDA with arPZQ will be documented and reported by using existing tools and established reporting pathways aligned with standard pharmacovigilance and safety guidelines of the national drug authorities. Based on routine program processes and forms, variables pertaining to drug logistics, training, drug distribution, passive pharmacovigilance and supervision will be collected in order to measure and generate real-world data related to feasibility, coverage and acceptability of selected platforms and strategies to inform future scale-up to district levels.

Assessments will take place before (to capture social mobilization and training activities) during and after the drug distribution to document the implementation process and evaluate experiences made by the different stakeholders (e.g. children, parents, community members, health workers, programme staff).

ELIGIBILITY:
* Living in the designated implementation area since at least 6 months
* Aged between 24 - 59 months
* Informed consent available
* No acute or chronic illness and/or inability to take oral medication
* No reported history of seizures
* No known allergic response to praziquantel

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Study population receiving intervention: All eligible preschool-aged children (2-5 years) from pre-selected study areas for small-scale implementation present at the day of the treatment campaign, will be accessed and treated with arpraziquantel by one of the two selected platforms depending on the assignment of the area.
  * Study population of post-distribution social science study: Subsamples of parents of preschool-aged children of the respective implementation areas, community stakeholders involved in social mobilization and distribution, health workers and programmatic staff involved in training, social mobilization and distribution.
Sampling Method: Non-Probability Sample
Enrollment: 18500 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Platform performance for arPZQ distribution | Documentation from 3 months before up to 12 weeks after the drug distribution
  Platform performance will be combined measure based on the coverage and feasibility measured by the following parameters and implementation outcome indicators:
  * Platform reach: Program reach and therapeutic coverage
  * Platform feasibility: Extent of changes to established procedures and requirements in terms of resources for social mobilization, training, drug logistics and drug delivery Feasibility will be assessed through quantitative and qualitative data on operational aspects
  * Platform acceptability/suitability: quantitative and qualitative feedback by stakeholders (health system & population perspective) assessed through Questionnaires & FGDs with parents and community stakeholders, KIIs and transect walks with health workers and programmatic supervision/monitoring tools and review meetings of implementers
  For the analysis and selection of a platform, a prioritization matrix will be developed which enables a triangulation and weighing of the above mentioned indicators.

SECONDARY OUTCOMES:
Effectiveness of social mobilization, communication and training | Documentation from 3 months before up to 12 weeks after the drug distribution
  The effectiveness of the advocacy, social mobilization and communication campaign will be measured as a combined measure by the following indicators:
  * Appropriateness of the tools (content, distribution channel, locations, timetable)
  * Acceptability of messages and motivation to access treatment
  * Coverage and scope of social mobilization
  * Feasibility in terms of equipment, personnel and timetable using questionnaires, FGDs, KIIs, non-participative observations through social scientists and routine monitoring and supervision tools as well as training knowledge assessment forms applied by the platforms and monitoring and evaluation teams.
  For the analysis and selection of a platform with regard to its social mobilization and communication effectiveness, a prioritization matrix will be developed which enables a triangulation and weighing of the above mentioned indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Steinmann, PhD PD, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (7):
- Côte d’Ivoire (3):
  - Programme National de Lutte Contre les Maladies Tropicales Négligées à Chimiothérapie Préventive (PNLMTN-CP), Ministère de la Santé, de l'Hygiène Publique et de la Couverture Maladie Universelle (MSHPCMU), Abidjan
  - Université Félix Hophouët-Boigny (UFHB), Département de sociologie, Abidjan
  - Université Félix Hophouët-Boigny (UFHB), UFR Biosciences, Abidjan
- Kenya (2):
  - African Institute for Health and Development (AIHD), Nairobi
  - Kenya Medical Research Institute (KEMRI), Eastern and Southern Africa Centre of International Parasite Control (ESACIPAC), Nairobi
- Uganda (2):
  - Makerere University, Department of Sociology and Anthropology, Kampala
  - Vector Borne & Neglected Tropical Disease Control Division, Ministry of Health, Kampala

IPD SHARING:
Plan to Share IPD: No
There are data sharing agreements (DTAs) between Swiss TPH, Côte d'Ivoire/Kenya/Uganda MoH, Felix Hophouët-Boigny University, Kenya Medical Research Institute and Makerere University in place. Likewise DTAs are in place between partners working on the social science study that is between Technical University München, the African Institute for Health & Development, Makerere University and Felix Hophouët-Boigny University. Data may be shared with other researchers upon request.